CLINICAL TRIAL: NCT02430896
Title: Neuropsychological, Genetic and Neuroimaging Markers and Treatment Response Predictors of Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Identification of Neuropsychological, Genetic and Neuroimaging Markers and Treatment Response Predictors of ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyo-Won Kim, Assistant professor, department of psychiatry, Asan Medical Center, Asan Medical Center
Other Study IDs: S2013-0373-0014
Record Dates: First submitted 2015-04-20; First posted 2015-04-30 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Neuropsychological; neuroimaging; genetic markers; treatment response predictor
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Atomoxetine Hydrochloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood sample for GWAS (Genome-Wide Association Study)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHD group: Children and adolescents who met the Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) diagnostic criteria for ADHD and needed pharmacotherapy. Subjects will be taking Methylphenidate or Atomoxetine for 52 weeks.
  Interventions: Drug: Methylphenidate (MPH); Drug: Atomoxetine
- Normal control group: Children and adolescents will be recruited by advertisement, and will be assigned to normal group if they do not meet the Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) diagnostic criteria for ADHD .

INTERVENTIONS:
Drug: Methylphenidate (MPH) — Subjects of ADHD group will be taking methylphenidate or atomoxetine for 52 weeks.
  Other Names: Metadate CD®; Concerta®; Medikinet Retard®
  Groups: ADHD group
Drug: Atomoxetine — Subjects of ADHD group will be taking methylphenidate or atomoxetine for 52 weeks.
  Other Names: Straterra®
  Groups: ADHD group

SUMMARY:
The objective of this study is to identification of neuropsychological, genetic and neuroimaging markers and treatment response predictors of attention-deficit/hyperactivity disorder (ADHD). Participants who take the standardized pharmacotherapy (methylphenidate or atomoxetine) for ADHD will be observed for 52 weeks. They will do several neuropsychological, neuroimaging and genetic tests at visit 1~6.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 6 and 12 years
2. met the Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) diagnostic criteria for ADHD and needed pharmacotherapy.
3. Informed consent

Exclusion Criteria:

1. presence of intellectual disability or learning disorder
2. past and/or current history of bipolar disorder or psychosis or substance use disorder
3. past and/or current history of pervasive developmental disorder, organic mental disorder or other neurological disorder
4. presence of sever suicidal ideation
5. presence of tic disorder or obsessive-compulsive disorder whose symptoms needed pharmacotherapy
6. presence of family history with Tourette's Syndrome
7. took medication with methylphenidate or atomoxetine with last 6 month (or more than 3 month)
8. presence of severe medical condition (ex. cardiologic, liver, kidney, pulmonary, glaucoma)
9. took alpha 2 adrenergic receptor agonist, antidepressant, antipsychotics, benzodiazepine, modafinil, antiepileptic drug or dietary supplement that have a influence on Central Nervous System (CNS).
10. presence of possibility with pregnancy
11. especially for neuroimaging,

    1. uncooperative with claustrophobia or body movement
    2. metal material inside body that can't take off

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Total 600 children and adolescents will be enrolled in this study. 500 patients in psychiatric outpatient will be enrolled. 100 persons of healthy volunteers will be recruited via advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Wide genome analysis regarding genetic polymorphisms as predictors of treatment response in Attention-Deficit/Hyperactivity Disorder(ADHD). | visit 1 (-week 8)
  Genome wide case-control association analysis will be operated with qualified phenotype and assigned intermittent phenotype.
Neuroimaging analysis as predictors of treatment response in Attention-Deficit/Hyperactivity Disorder(ADHD). | visit 1 (-week 8)
  Thickness of cortex, anatomical relation will be compared with 3 tesla MRI. In addition, brain circuit for delayed aversion, delayed frustration, time processing and resting state.
Drug effectiveness is assessed using ADHD rating scale, CGI -S (Clinical Global Impression - Severity scale) and CGI-I (Clinical Global Impression - Improvement scale). | visit 1 (-week 8)
Neuropsychological markers as the treatment response predictable factor of ADHD using a complex neuropsychological test consisting of SSRT, delayed aversion, delayed frustration, time processing, ATA | visit 1 (-week 8)
  Using a complex neuropsychological test consisting of The stop-signal reaction time (SSRT) task, delayed aversion, delayed frustration, time processing, Advanced tets of Attention (ATA).
Comorbidity assessment using a composite measure consisting of K-PRC, C-SSRS, TCGI, and DCDQ | visit1 (-week 8)
  It is assessed using a composite measure consisting of Korean Personality Rating Scale for Children (K-PRC), Columbia Suicide Severity Rating Scale (C-SSRS), The Tic Severity Scale (TCGI), and The Developmental Coordination Disorder Questionnaire (DCDQ).

OTHER OUTCOMES:
Change from baseline in treatment response effectiveness of pharmacotherapy at week12 | visit 3 (week12)
  Drug effectiveness is assessed using ADHD rating scale, CGI -S (Clinical Global Impression - Severity scale) and CGI-I (Clinical Global Impression - Improvement scale).
Change from baseline in treatment response effectiveness of pharmacotherapy at week 24 | visit 4 (week 24)
  Drug effectiveness is assessed using ADHD rating scale, CGI -S (Clinical Global Impression - Severity scale) and CGI-I (Clinical Global Impression - Improvement scale).
Change from baseline in treatment response effectiveness of pharmacotherapy at week 36 | visit 5 (week 36)
  Drug effectiveness is assessed using ADHD rating scale, CGI -S (Clinical Global Impression - Severity scale) and CGI-I (Clinical Global Impression - Improvement scale).
Change from baseline in treatment response effectiveness of pharmacotherapy at week 52 | visit 6 (week 52)
  Drug effectiveness is assessed using ADHD rating scale, CGI -S (Clinical Global Impression - Severity scale) and CGI-I (Clinical Global Impression - Improvement scale).
Change from baseline in neuropsychological markers as the treatment response predictable factor of ADHD using a complex neuropsychological test consisting of SSRT, delayed aversion, delayed frustration, time processing, ATA at week 12 | visit 3 (week 12)
  Using a complex neuropsychological test consisting of The stop-signal reaction time (SSRT) task, delayed aversion, delayed frustration, time processing, Advanced tets of Attention (ATA).
Change from baseline in neuropsychological markers as the treatment response predictable factor of ADHD using a complex neuropsychological test consisting of SSRT, delayed aversion, delayed frustration, time processing, ATA at week 52 | visit 6 (week 52)
  Using a complex neuropsychological test consisting of The stop-signal reaction time (SSRT) task, delayed aversion, delayed frustration, time processing, Advanced tets of Attention (ATA).
Occurrence of comorbidity from baseline in assessment using a composite measure consisting of K-PRC, C-SSRS, TCGI, and DCDQ at week 12 | visit 3 (week 12)
  It is assessed using a composite measure consisting of Korean Personality Rating Scale for Children (K-PRC), Columbia Suicide Severity Rating Scale (C-SSRS), The Tic Severity Scale (TCGI), and The Developmental Coordination Disorder Questionnaire (DCDQ).
Occurrence of comorbidity from baseline in assessment using a composite measure consisting of K-PRC, C-SSRS, TCGI, and DCDQ at week 52 | visit 6 (week 52)
  It is assessed using a composite measure consisting of Korean Personality Rating Scale for Children (K-PRC), Columbia Suicide Severity Rating Scale (C-SSRS), The Tic Severity Scale (TCGI), and The Developmental Coordination Disorder Questionnaire (DCDQ).

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Won Kim, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No